CLINICAL TRIAL: NCT04892732
Title: Replication of the D58 Asthma Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-D58
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Budesonide: Reference Group
  Interventions: Drug: Budesonide
- Budesonide-formoterol: Exposure Group
  Interventions: Drug: Budesonide-Formoterol

INTERVENTIONS:
Drug: Budesonide — Budesonide dispensing claim is used as the reference group.
  Groups: Budesonide
Drug: Budesonide-Formoterol — Budesonide-Formoterol dispensing claim is used as the exposure group.
  Groups: Budesonide-formoterol

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Criteria:

Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates:

Budesonide-formoterol was approved by FDA on July 21, 2006 for management of asthma. The initial eligible cohort entry date was the first date after July 21, 2006 for both the databases investigated (IBM MarketScan, Optum CDM). The last date eligible as cohort entry date was the end of available data for IBM MarketScan and Optum CDM. The following eligible cohort entry dates were included:

* IBM MarketScan: July 21, 2006 - December 31, 2018 (end of available data)
* Optum CDM: July 21, 2006 - June 30, 2020 (end of available data)

Inclusion Criteria:

* ≥12 years of age
* Documented clinical diagnosis of asthma for ≥1 year prior to randomization
* History of at least one asthma exacerbation in the previous year (but none in the 4 weeks prior to randomization. An asthma exacerbation was defined as an event requiring treatment with systemic corticosteroids or requiring hospitalization (i.e. an inpatient stay or >24-hour stay in the observation area of an emergency room or local equivalent)
* Receiving either:

  1. A stable dose of ICS alone or in combination with a LABA, leukotriene receptor antagonist or other maintenance therapy/therapies for ≥4 weeks prior to randomization (any patient maintained on a stable high-dose ICS with or without a LABA or LTRA or other maintenance therapy/therapies was required to have an ACQ6 total score of <1.5 at screening) OR
  2. A stable dose of LTRA or xanthine monotherapy (for ≥4 weeks prior to randomization) or daily SABA (in the 4 weeks before randomization but ≤8 puffs a day on two consecutive days, or ≥25 puffs in one day, in the 7 days prior to screening). Patients on LTRAs, xanthines, or daily SABA, were eligible only if they recorded an ACQ6 total score of ≥1.5, and in the investigator's clinical judgment, the patient's asthma severity could have justified treatment with ICS or ICS/LABA combination

Exclusion Criteria:

* A history of life-threatening asthma (defined as an asthma episode that required intubation and/or was associated with hypercapnia requiring non-invasive ventilatory support)
* One of the following:

  1. Any asthma exacerbation requiring systemic corticosteroids within 4 weeks prior to randomization OR
  2. >4 separate exacerbations OR
  3. >2 hospitalizations (an inpatient stay or >24- hour stay in the observation area of an emergency room or local equivalent) due to asthma in the previous year
* Received systemic corticosteroids for any reason in the 4 weeks prior to randomization
* Had an ongoing asthma exacerbation requiring systemic corticosteroids
* Concurrent respiratory disease (chronic obstructive pulmonary disease, chronic bronchitis, emphysema, idiopathic pulmonary fibrosis, bronchiectasis, and/or any pulmonary disease)
* A smoking history of >10 pack-years
* Respiratory infection or other viral/bacterial illness
* Pregnancy (current/planned) and lactation
* Malignancy (with the exception of basal cell carcinoma) within the 5 years prior to study commencement
* Omalizumab or any other monoclonal/polyclonal antibody use in the 6 months prior to randomization
* Concomitant β-blocker use
* Drug/alcohol abuse

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort design comparing budesonide-formoterol versus budesonide alone. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of budesonide-formoterol or budesonide.
Sampling Method: Non-Probability Sample
Enrollment: 66581 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
First serious asthma-related event | Through study completion (a median of 88-116 days)
  A composite of adjudicated death, intubation, and hospitalization

SECONDARY OUTCOMES:
Asthma-related hospitalization | Through study completion (a median of 88-116 days)
Asthma-related intubation | Through study completion (a median of 88-116 days)
Asthma-related death | Through study completion (a median of 88-116 days)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT04892732/Prot_SAP_001.pdf